CLINICAL TRIAL: NCT01816191
Title: An Open-Label, Single- and Multi-Dose Pharmacokinetic (PK) Study of Oral Diltiazem and Topical Diltiazem Hydrochloride
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ventrus Biosciences, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VEN307-PK-001
Record Dates: First submitted 2013-03-13; First posted 2013-03-22 (Estimated); Last update posted 2013-08-21 (Estimated); Status verified 2013-07

CONDITIONS: Adult Subjects With Anal Fissures.
MeSH Terms: interventions — Diltiazem

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Diltiazem Hydrochloride (Experimental): Topical cream and oral pill
  Interventions: Drug: Diltiazem Hydrochloride Cream and Oral Diltiazem

INTERVENTIONS:
Drug: Diltiazem Hydrochloride Cream and Oral Diltiazem

SUMMARY:
The study is a single-center, open-label, safety and pharmacokinetic study in12 adult subjects with Anal Fissures. Subjects will be screened to determine eligibility within 7 days of treatment. There will be three parts to the study and all subjects will participate in each part.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with evidence of a circumscribed anal fissure, with induration at the edges.
* Any female of non-childbearing potential who:

  a) has had a hysterectomy, b) has had a bilateral oophorectomy, c) has had a bilateral tubal ligation or d) is post-menopausal (demonstration of total cessation of menses for ≥ 1 year from the date of the screening visit).
* Any female of child bearing potential must agree to use at least one form of contraception(may be a barrier method), during the full duration of the study.
* Able to communicate adequately with the investigator and to comply with the requirements for the entire study.
* Capable of and freely willing to provide written informed consent prior to participating in the study.

Exclusion Criteria:

* Unwilling to have visual or medical examination of the Anal Fissure.
* More than 1 Anal Fissure.
* Subjects with Anal Fissure associated with or caused by other conditions, including but not limited to: drug-induced, trauma, HIV infection, fistula-in-ano, inflammatory bowel disease, perianal sepsis or malignancy.
* Unwilling to stop all other concomitant topical preparations applied in and around the anus from Day -1 through end of the study.
* Use of sitz bath from signing of ICF (Informed Consent Form) to end of study.
* Use of anesthetics from signing the ICF to end of study.
* Subfissure injection of botulinum toxin in the 3 months prior to signing the ICF.
* Known sensitivity to investigational product(s) or calcium channel blockers.
* Active treatment with anti-viral therapies for HIV (e.g. indinavir, nelfinivir,ritonavir).

  10. Treatment with any prohibited medications within 14 days prior to signing the ICF:
  * Cytochrome P450 (CYP450) inhibitors and inducers
  * Cytochrome P3A4 (CYP3A4) substrates, inhibitors, and inducers
  * Benzodiazepines
  * β-adrenoceptor antagonists (Beta-Blockers)
  * Calcium channel blockers
  * Digoxin
  * Investigational agents
  * Opioids
* Following concomitant disease state:

  * Sick sinus syndrome except in the presence of a functioning ventricular pacemaker.
  * Second-or third-degree Atrioventricular block except in the presence of a functioning ventricular pacemaker.
  * Hypotension (less than 90 mm Hg systolic).
  * Acute myocardial infarction and pulmonary congestion documented by x-ray.
  * History of clinically significant renal disease.
  * History of clinically significant Alzheimer's or Parkinson's disease.
  * History of clinically significant hepatic disease.
  * Current infection treated with a macrolide antibiotic.
  * Clinical evidence or history of fecal incontinence.
  * Clinical evidence or history of anal fistula.
  * Clinical evidence or history of anal abscess.
  * History of inflammatory bowel disease (e.g. Crohn's disease, Ulcerative Colitis).
  * History of any prior anal or rectal surgery including but not limited to: lateral sphincterotomy and anal stretch.
* History of radiation therapy to the pelvis.
* Fixed anal stenosis/fibrosis.
* Major organ transplant.
* Any clinically significant laboratory abnormalities during screening.
* BMI > 40 kg/m2.
* Malignancy within 5 years prior to randomization (with the exception of treated basal cell/squamous cell carcinoma of the skin).
* Any disease or prior/planned surgery that may interfere with the subject successfully completing the study.
* Currently using narcotic(s) chronically.
* Breast-feeding females.
* Employees, family members, or students of the investigator or clinical site.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2013-02; Primary Completion 2013-07 (Actual); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
Single and multiple dose Pharmacokinetic parameters | up to 6 months after enrollment begins
  Single- and multiple-dose PK parameters for topical DTZ and single-dose PK parameters for oral DTZ including AUC(0-t), AUC(0-∞), Cmax, tmax, t1/2 and CL/F. PK parameters for DTZ, and its two metabolites (N-desmethylditiazem and O-desacetyldiltiazem) will be presented in Data Listings and summarized by Day (Study Day 1, 7 and 14). Descriptive statistics will include n, mean, SD, %CV, geometric mean,median, minimum, and maximum.

SECONDARY OUTCOMES:
Safety as determined by nature, severity and relationship of adverse events, clinical labs, physical exam findings, vital signs and Electrocardiogram | Up to 6 months after enrollment begins
  Adverse events, physical examination findings, vital sign measurements, ECG results, and clinical laboratory data will be reviewed and summarized to evaluate the safety profile of topical DTZ cream and oral DTZ. Safety data will be summarized by study time point, and by change from Baseline using descriptive statistics as appropriate. Data listings will also be provided.

CONTACTS AND LOCATIONS:
Locations (1):
- Wake Research Associates, Raleigh, North Carolina, United States